CLINICAL TRIAL: NCT02527408
Title: Wearable Technology for Hospital Inpatients
Acronym: WEARIT-IN
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. David Maslove, Assistant Professor, Queen's University
Other Study IDs: DMED-1818-15
Record Dates: First submitted 2015-08-13; First posted 2015-08-19 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Heart Rate Monitoring

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will address the feasibility of using wrist-worn fitness trackers to monitor hospital inpatients. The study is being conducted in the Intensive Care Unit where patients are closely monitored, in order to provide gold standard measurements of heart rate, and accurate estimates of sleep quality.

DETAILED DESCRIPTION:
Overall Hypothesis:

The use of wearable personal fitness trackers to monitor physiologic signals in hospital inpatients is feasible, reliable, secure, and cost effective.

Specific Objectives:

1. To evaluate the feasibility of applying a wrist-worn personal fitness tracker to hospital inpatients for the purpose of monitoring heart rate and sleep quality during the night.
2. To determine the accuracy and completeness of high-frequency heart rate measurements recorded from personal fitness trackers in hospital inpatients.
3. To compare measurements of sleep quality generated by personal fitness trackers with clinical assessments by nursing staff among hospital inpatients.
4. To develop a workflow and data analysis pipeline for downloading, storing, analyzing, and visualizing data generated by personal fitness trackers worn by hospital inpatients.
5. To evaluate the feasibility of a larger prospective multicenter trial examining the utility of personal fitness trackers among hospital inpatients, including recruitment rates, inclusion/exclusion criteria, data management protocols, and outcomes measures.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age > 18 years)
2. Spontaneously breathing (i.e. no invasive or non-invasive mechanical ventilation, with the exception of nocturnal non-invasive ventilation at stable home settings)
3. Cardiac telemetry and/or continuous SpO2 monitoring in place

Exclusion Criteria:

1. Continuous sedation or analgesia
2. Known upper extremity deep venous thrombosis
3. Dialysis fistula
4. Radial arterial line in the non-dominant arm
5. Peripherally inserted central venous catheter in the non-dominant arm
6. Severe upper extremity trauma or fracture
7. History of upper extremity amputation
8. Skin breakdown at application site
9. Contact precautions (methicillin resistant Staph aureus, C. difficile, vancomycin resistant Enterococcus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Heart rate accuracy | 6 months
  Percentage of heart rate measurements that are within 5 beats per minute of telemetry reading

SECONDARY OUTCOMES:
Agreement with sleep quality questionnaire | 6 months
  Correlation between Fitbit derived sleep quality score, and the Richards-Campbell Sleep Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Maslove, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Kroll RR, McKenzie ED, Boyd JG, Sheth P, Howes D, Wood M, Maslove DM; WEARable Information Technology for hospital INpatients (WEARIT-IN) study group. Use of wearable devices for post-discharge monitoring of ICU patients: a feasibility study. J Intensive Care. 2017 Nov 21;5:64. doi: 10.1186/s40560-017-0261-9. eCollection 2017. PMID 29201377
- [Derived] Kroll RR, Boyd JG, Maslove DM. Accuracy of a Wrist-Worn Wearable Device for Monitoring Heart Rates in Hospital Inpatients: A Prospective Observational Study. J Med Internet Res. 2016 Sep 20;18(9):e253. doi: 10.2196/jmir.6025. PMID 27651304